CLINICAL TRIAL: NCT04470752
Title: Capsaicin for Post-stroke Dysphagia
Acronym: CADYS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georg Kägi, MD (Other)
Collaborators: Cantonal Hospital of Aarau, Switzerland (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Georg Kägi, MD, Senior Physician and Head of the Stroke Center, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BASEC 2020-01362; 08.011 (Other: CTU Kantonsspital St. Gallen)
Record Dates: First submitted 2020-06-02; First posted 2020-07-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Dysphagia, Late Effect of Stroke
Keywords: Dysphagia; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Capsaicin; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both study drug and Placebo have identical packaging (brown glass bottle) and labeling (Capsaicin or Placebo). Both use the same liquid suspension, same colour, and consistency..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): InOrpha solution/ml, three times daily with meals for the Treatment period, 7 or 30 days.
  Interventions: Drug: InOrpha Solution
- Capsaicin (Experimental): InOrpha solution plus 1 mcg Capsaicin/ml, three times daily with meals for the Treatment period of 7 or 30 days.
  Interventions: Drug: Capsaicin 1% oral solution

INTERVENTIONS:
Drug: Capsaicin 1% oral solution — Capsaicin 1.0 micrograms/ml
  Arms: Capsaicin
Drug: InOrpha Solution — glycerol based suspension vehicle
  Arms: Placebo

SUMMARY:
Randomised, double blind, Phase 2 Trial to evaluate the efficacy of oral Capsaicin in patients with post-stroke dysphagia in the (sub-)acute setting.

DETAILED DESCRIPTION:
After inclusion and the assessment of the swallowing function (PRESS, PAS, FOIS, FEES) patients will be randomised 1:1 to receive 1mcg Capsaicin or Placebo. Oral treatment will be applied 3 times daily either during meals or during regular swallowing tests/trainings accompanied by a Speech Language Pathologist. After re-assessment of the dysphagia after 7 days, patients with persistent dysphagia and applicable for further treatment will be treated for another 23 days with a final clinical swallowing evaluation after a total of 30 days. A Patient Medication Diary will used during the Duration of the Trial to capture compliance.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic Stroke
* Impairment of oral intake with FOIS ≤ 4
* Magnetic Resonance Imaging of the brain or CT scan with the finding of a subacute ischemic stroke
* Informed Consent within 48 hours after admission, following initial swallowing assessment

Exclusion Criteria:

* Diagnosis other than ischemic stroke
* Late patient admission >48 hours after stroke onset
* Impairment of functional oral intake scale ≥ 5
* FEES >72h after admission
* PAS <2
* Pre-existing dysphagia
* Dysphagia due to other cause
* No evidence of stroke on imaging
* Recurrent stroke = at least one stroke in the course of the study apart from the index stroke
* Age <18 years
* Current drug abuse
* Amphetamine or amphetamine-like Medication
* Regular oral treatment with chilli pepper extract
* Allergies or known adverse reactions to the consumption of chilli pepper or capsaicin
* Personality disorder
* Severe dementia or delirium
* Other reasons according to physician/investigator because of which the patient cannot participate in the study (not suitable for treatment or examinations)
* withdrawal of consent by participant at any time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Penetration Aspiration Scale (PAS) score | 7 days after randomisation
  the between-group difference of the Penetration Aspiration Scale (PAS) assessed with functional endoscopic evaluation of swallowing (FEES) 7 days after admission.

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) score | at day 7 and 30 post admission
  Between group differences (capsaicin / placebo) of Functional Oral Intake Scale (FOIS)
days of nasogastric tube feeding | from randomisation until day 30
  Between group differences (capsaicin / placebo) of days of nasogastric tube feedings
number of patients with Percutaneous endoscopic gastrostomy (PEG) tube placement | from randomisation until day 30
  Between group differences (capsaicin / Placebo) of number of patients with PEG tube placement
number of patients with aspiration pneumonia | from randomisation until day 30
  Between group differences (capsaicin / Placebo) of number of patients with aspiration pneumonia
Swallowing quality of life questionnaire (Swal-QoL) score | from randomisation until day 30
  Between group differences (capsaicin / Placebo) of Swallowing quality of life questionnaire (Swal-QoL)
Latency of the Swallowing reflex | from randomisation until day 30
  Between group differences (capsaicin / Placebo) of Latency of the Swallowing reflex
modified Ranking Scale (mRS) score | from randomisation until day 30
  Between group differences (capsaicin / Placebo) of modified Ranking Scale (mRS)
Change of Penetration Aspiration Scale (PAS) and/or Functional Oral Intake Score (FOIS) with supratentorial stroke | after 7 and 30 days post admission
  admission of patients with and without sensory deficits (only supratentorial strokes)
Change of Penetration Aspiration Scale (PAS) and/or Functional Oral Intake with supra-infratentorial stroke | after 7 and 30 days post admission
  of patients with stroke localisation with respect to supra-infratentorial localisation and involvement of sensory/motor swallowing cortex with its connections

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | 30 days post admission
  Potential harm will be assessed by comparing between-group differences (verum/placebo) of hypothermia and other (serious) adverse events which are not known yet, but will be collected systemically during this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Georg kägi, Dr. med., Principal Investigator — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We plan to upload the study protocol after trial completion
Supporting Information: Study Protocol
Time Frame: after Trial completion indefinitely

REFERENCES:
- See also: PRESS App — https://play.google.com/store/apps/details?id=ch.kssg.press&hl=en_US